CLINICAL TRIAL: NCT00787865
Title: Diffusion Tensor Imaging (DTI) as a Tool to Identify Infants With Krabbe Disease in Urgent Need of Treatment
Brief Title: Diffusion Tensor Imaging (DTI) in Infants With Krabbe Disease
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Deepa Soundara Rajan, Assistant Professor, University of Pittsburgh
Other Study IDs: STUDY20020124; R01NS061965 (NIH)
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Krabbe Disease
Keywords: Diffusion Tensor Imaging; DTI; Newborn; Krabbe Disease; Motor Development; Motor Disability
MeSH Terms: conditions — Leukodystrophy, Globoid Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (4):
- Krabbe Disease: Children with infantile Krabbe disease
- Low Enzyme/No Krabbe Disease: Children without disease who have low enzyme levels
- Control: Children with no disease and normal enzyme levels
- Motor Disability: Children at risk of developing motor disability

SUMMARY:
This study is designed to learn about early brain development in children with Krabbe disease, and to use diffusion tensor imaging as an early diagnostic tool to identify newborns at risk for the disease.

DETAILED DESCRIPTION:
This study is designed to learn about early brain development in children with Krabbe disease and to use diffusion tensor imaging (DTI) as an early diagnostic tool to differentiate children with infantile Krabbe disease from newborns who are disease free but have very low enzyme levels. Additionally, this study will determine how certain structures in the brain will develop over 24 months in children with infantile Krabbe disease and those without disease who have low enzyme levels. This study will also reveal information about the learning and motor development of children, and will help researchers predict outcomes after treatment.

Krabbe disease is a rare, childhood neurodegenerative disorder caused by galactocerebrosidase deficiency. It results in rapid demyelination, progressive spasticity, mental deterioration, blindness, deafness, seizures, and death. Based on previously published findings, treatment with unrelated umbilical cord blood transplantation is now standard for Krabbe disease, provided that the treatment occurs within the first weeks of life and before symptoms appear.

Once newborns are identified through population screening, there is no objective measure to predict if the baby will develop the most frequent rapidly progressive infantile forms of Krabbe or have a slower juvenile or adult form. Phenotype and genotype correlations are not possible because there are more than 150 mutations that can cause the disease and many polymorphisms in the normal population that affect the enzyme level.

There is an urgent clinical need to develop a predictive measure. To date, there are no available tools to classify infants into the infantile versus later forms. New advances in neuroimaging techniques have enabled scientists to quantify changes in brain growth and myelination early in life and before disease symptoms develop.

Knowledge from this study will help identify the window of opportunity for early intervention and treatment to prevent severe disability, and may lead to better treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Positive newborn screening test (low galactocerebrosidase)
2. Infantile Krabbe Disease diagnosed by confirmatory low levels of residual enzyme by Dr. Wenger's Lysosmal Storage Diseases laboratory at Jefferson's Medical College (contracted by New York State) and/or carrier status established because of family history of Krabbe Disease. Patients have to be less than 6 weeks old at the time of the first assessment
3. Children at risk of developing motor disability

Exclusion Criteria:

1. Diagnosis or physical signs of known genetic conditions or syndromes, serious medical or neurological conditions affecting growth and development (e.g., seizure disorder, diabetes, congenital heart disease) or sensory impairments such as vision or hearing loss
2. Children who may have suffered serious perinatal brain damage, children with birth weights less than 2000 grams and/or gestational ages of less than 34 weeks, or those with a history of intraventricular hemorrhage
3. Children who may have a contraindication for MRI (pacemaker, vascular stents, metallic ear tubes, other metal implants or braces).

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with a low levels of galactocerebrosidase, a family history of Krabbe disease or has been diagnosed with Krabbe disease, or is a child at risk of developing motor disability. Newborn screening State of New York and newborns with low enzyme.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-04; Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Diffusion tensor imaging (DTI) of corticospinal tracts | at birth, 1 year and 2 years of age

SECONDARY OUTCOMES:
Motor development at birth, 1 year and 2 years of age | at birth, 1 year and 2 years of age
Analysis of DTI-Fractional Diffusion Anisotropy (FA) values of corticospinal tracts of newborns | at age (newborn-6 weeks), 12-months and 24-months

CONTACTS AND LOCATIONS:
Overall Officials: Deepa S Rajan, MD, Principal Investigator — University of Pittsburgh School of Medicine, Children's Hospital of Pittsburgh-UPMC
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Escolar ML, Poe MD, Provenzale JM, Richards KC, Allison J, Wood S, Wenger DA, Pietryga D, Wall D, Champagne M, Morse R, Krivit W, Kurtzberg J. Transplantation of umbilical-cord blood in babies with infantile Krabbe's disease. N Engl J Med. 2005 May 19;352(20):2069-81. doi: 10.1056/NEJMoa042604. PMID 15901860
- [Background] Provenzale JM, Escolar M, Kurtzberg J. Quantitative analysis of diffusion tensor imaging data in serial assessment of Krabbe disease. Ann N Y Acad Sci. 2005 Dec;1064:220-9. doi: 10.1196/annals.1340.040. PMID 16394159
- See also: Information about the Program for the Study of Neurodevelopment in Rare Disorders — https://www.chp.edu/our-services/ndrd